CLINICAL TRIAL: NCT05383352
Title: A Phase I, Randomised, Open-Label, Single-Dose, Two-Treatment, Two-Way Crossover, Two-Stage Study to Evaluate the Bioequivalence of Onivyde (Irinotecan Liposome Injection) Manufactured at Two Different Sites Administered in Combination With Anti-Cancer Agents in Adult Participants With Metastatic Pancreatic Adenocarcinoma
Brief Title: A Study to Compare Onivyde Manufactured at Two Different Production Sites in Adult Participants With Advanced Cancer in the Pancreas
Acronym: SIRACUSA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D-FR-60010-015; 2021-003264-26 (EudraCT Number)
Record Dates: First submitted 2022-05-03; First posted 2022-05-20 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Metastatic Pancreatic Adenocarcinoma
MeSH Terms: interventions — irinotecan sucrosofate; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sequence RT: Reference Product followed by Test Product (Experimental): Cycle 1 (Crossover Phase) Day 1: One dose Onivyde® Reference product + 5-FU/LV.
  Cycle 1 (Crossover Phase) Day 15: One dose Onivyde Test product + 5-FU/LV
  Cycle 2 Onwards (Extension Phase): Participants who choose to continue treatment after Cycle 1 will receive Onivyde® Reference product on Day 1 and Day 15 of every 28-day cycle in combination with 5-FU/LV
  Interventions: Drug: Irinotecan liposome injection; Drug: Folinic Acid; Drug: 5-Fluorouracil
- Sequence TR: Test Product followed by Reference Product (Experimental): Cycle 1 (Crossover Phase) Day 1: One dose Onivyde Test product + 5-FU/LV.
  Cycle 1 (Crossover Phase) Day 15: One dose Onivyde® Reference product + 5-FU/LV.
  Cycle 2 Onwards (Extension Phase): Participants who choose to continue treatment after Cycle 1 will receive Onivyde® Reference product on Day 1 and Day 15 of every 28-day cycle in combination with 5-FU/LV.
  Interventions: Drug: Irinotecan liposome injection; Drug: Folinic Acid; Drug: 5-Fluorouracil

INTERVENTIONS:
Drug: Irinotecan liposome injection — Onivyde 70 mg/m2 intravenously over 90 minutes on Cycle 1 Day 1 (Crossover Phase) and from cycle 2 onwards on Day 1 and Day 15 of every 28-day cycle (Extension Phase)
  Other Names: Onivyde® Reference product
  Arms: Sequence RT: Reference Product followed by Test Product
Drug: Irinotecan liposome injection — Onivyde 70 mg/m2 intravenously over 90 minutes on Cycle 1 Day 15 (Crossover Phase)
  Other Names: Onivyde Test product
  Arms: Sequence RT: Reference Product followed by Test Product
Drug: Irinotecan liposome injection — Onivyde 70 mg/m2 intravenously over 90 minutes on Cycle 1 Day 1 (Crossover Phase)
  Other Names: Onivyde Test product
  Arms: Sequence TR: Test Product followed by Reference Product
Drug: Irinotecan liposome injection — Onivyde 70 mg/m2 intravenously over 90 minutes on Cycle 1 Day 15 (Crossover Phase) and from cycle 2 onwards on Day 1 and Day 15 of every 28-day cycle (Extension Phase)
  Other Names: Onivyde® Reference product
  Arms: Sequence TR: Test Product followed by Reference Product
Drug: Folinic Acid — LV 400 mg/m2 intravenously over 30 minutes, on Day 1 and Day 15 of every 28-day cycle
  Other Names: Leucovorin (LV)
Drug: 5-Fluorouracil — 5-FU 2,400 mg/m2 intravenously over 46 hours, on Day 1 and Day 15 every 28-day cycle
  Other Names: 5-FU

SUMMARY:
The aim of this study is to compare Onivyde manufactured at two different production sites in adult participants with advanced cancer in the pancreas.

Adult participants with metastatic pancreatic adenocarcinoma will receive Test Product (TP) and Reference Product (RP) Onivyde in line with its approved indication. The order in which they receive them depends on the group to which they are randomly assigned, this will be referred to as the crossover phase.

The average study duration for each participant until end of crossover phase is estimated to be approximately 3 months. After completion of the crossover phase, participants who in the opinion of the investigator will benefit from the treatment will be offered to enter the extension phase where they will receive the commercial Onivyde (RP) until disease progression, withdrawal, unacceptable toxicity or death. Metastatic pancreatic adenocarcinoma is a cancer that has spread (metastasized) beyond the area of the pancreas to other organs of the body.

Onivyde is approved for the treatment of metastatic adenocarcinoma of the pancreas after disease progression following gemcitabine-based therapy, in combination with 5-fluorouracil (5-FU) and leucovorin (LV).

ELIGIBILITY:
Inclusion Criteria :

* Participant must be ≥18 years of age at the time of signing the informed consent.
* Participants who have histological or cytologically confirmed adenocarcinoma of the pancreas.
* Participants with an initial diagnosis of progressive metastatic disease
* Participants with a confirmed diagnosis of metastatic adenocarcinoma of the pancreas with disease progression following gemcitabine-based therapy.
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤1
* Adequate haematological parameters
* Adequate hepatic function
* Adequate renal function
* Adequate coagulation
* No clinically significant abnormalities in urinalysis results
* Electrocardiogram (ECG) without any clinically significant findings
* Participants known to be infected with controlled human immunodeficiency virus (HIV)
* Male and female participants: Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies
* Capable of giving signed informed consent

Exclusion Criteria :

* Have only localised advanced disease.
* History of any second malignancy in the last 2 years.
* Known history of central nervous system metastases
* Clinically significant gastrointestinal disorder including hepatic disorders, bleeding, inflammation, occlusion, diarrhoea >Grade 1, malabsorption syndrome, ulcerative colitis, inflammatory bowel disease or partial bowel obstruction.
* Concurrent illnesses that would be a relative contraindication to trial participation such as active cardiac or liver disease
* Active infection or an unexplained fever >38.5°C on the first scheduled day of dosing
* Neuroendocrine tumour (carcinoid, islet cell) or acinar pancreatic carcinoma
* History of interstitial lung disease, history of slowly progressive dyspnoea and unproductive cough, sarcoidosis, silicosis, idiopathic pulmonary fibrosis, pulmonary hypersensitivity pneumonitis or multiple allergies.
* Exposure to a non-liposomal irinotecan or SN-38 based regimen within 4 weeks prior to randomisation, or exposure to Onivyde or other irinotecan based liposomal products within 6 weeks prior to randomisation
* Major surgery, other than diagnostic surgery, within 4 weeks prior to randomisation
* Participants who have received a live vaccine within 4 weeks prior to randomisation.
* Use of strong CYP3A inhibitors or inducers, or strong inhibitors of UGT1A1.
* Investigational therapy administered within 4 weeks, or within a time interval less than at least 5 half-lives of the investigational agent, whichever is longer, prior to study intervention on Cycle 1 Day 1
* Known low or absent dihydropyrimidine dehydrogenase (DPD) activity.
* Homozygous for the UGT1A1*28 allele.
* Known hypersensitivity to any of the components of Onivyde injection, other liposomal products, or any components of 5-FU, or LV
* Presence of any contraindications outlined in the Contraindications or Warnings and Precautions sections of the IB for Onivyde, or in the prescribing information for 5-FU or LV.
* Participants who, in the opinion of the investigator, have symptoms or signs suggestive of clinically unacceptable deterioration of the primary disease at the time of screening
* Any other medical or social condition deemed by the investigator to be likely to interfere with a participant's ability to sign informed consent, cooperate and participate in the study, or interfere with the interpretation of the results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2024-05-27 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Maximum (peak) plasma drug concentration (Cmax) of encapsulated irinotecan for Test relative to and Reference product | Crossover Phase (From Cycle 1 Day 1 to Day 28 and Cycle 1 Day 29 (pre-dose))
Area under the plasma concentration-time curve from time 0 to time t (AUC(0-t) of encapsulated irinotecan for Test relative to Reference product | Crossover Phase (From Cycle 1 Day 1 to Day 28 and Cycle 1 Day 29 (pre-dose))
Area under the plasma concentration-time curve from time 0 to infinity (AUC(0-∞) of encapsulated irinotecan for Test relative to Reference product | Crossover Phase (From Cycle 1 Day 1 to Day 28 and Cycle 1 Day 29 (pre-dose))

SECONDARY OUTCOMES:
Maximum (peak) plasma drug concentration (Cmax) of total irinotecan for Test relative to Reference product | Crossover Phase (From Cycle 1 Day 1 to Day 28 and Cycle 1 Day 29 (pre-dose))
Area under the plasma concentration-time curve from time 0 to time t (AUC(0-t)) of total irinotecan for Test relative to Reference product | Crossover Phase (From Cycle 1 Day 1 to Day 28 and Cycle 1 Day 29 (pre-dose))
Area under the plasma concentration-time curve from time 0 to infinity (AUC(0-∞)) of total irinotecan for Test relative to Reference product | Crossover Phase (From Cycle 1 Day 1 to Day 28 and Cycle 1 Day 29 (pre-dose))
Time to maximum plasma concentration (Tmax) of encapsulated and total irinotecan over 15-days for each Test and Reference products | Crossover Phase (From Cycle 1 Day 1 to Day 28 and Cycle 1 Day 29 (pre-dose))
Apparent clearance of drug from plasma (CL) of encapsulated and total irinotecan for Test and Reference products | Crossover Phase (From Cycle 1 Day 1 to Day 28 and Cycle 1 Day 29 (pre-dose))
Apparent volume of distribution (VZ) of encapsulated and total irinotecan for Test and Reference products | Crossover Phase (From Cycle 1 Day 1 to Day 28 and Cycle 1 Day 29 (pre-dose))
Terminal half-life (t1/2) of encapsulated and total irinotecan for Test and Reference products | Crossover Phase (From Cycle 1 Day 1 to Day 28 and Cycle 1 Day 29 (pre-dose))
Apparent terminal elimination rate constant (λZ) of encapsulated and total irinotecan for Test and Reference products | Crossover Phase (From Cycle 1 Day 1 to Day 28 and Cycle 1 Day 29 (pre-dose))
Percentage of participants with treatment-emergent adverse events (TEAEs) treatment-related leading to discontinuations, or to death | Crossover Phase (From Cycle 1 Day 1 to Day 28 and Cycle 1 Day 29 (pre-dose))
  Including treatment-emergent serious adverse events
Percentage of participants with clinically significant abnormal values | Crossover Phase (From Cycle 1 Day 1 to Day 28 and Cycle 1 Day 29 (pre-dose))
  It includes clinically significant abnormal laboratory results, physical examination findings, Electrocardiogram (ECG) and vital signs

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (36):
- Australia (2):
  - Flinders Medical Centre, Bedford Park
  - Peninsula and Southeast Oncology - Frankston Private Hospital, Frankston
- France (5):
  - Institut BERGONIE Centre de Lutte Contre le Cancer, Bordeaux
  - Centre GEORGES FRANÇOIS LECLERC, Dijon
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Chu La Miletrie, Poitiers
  - Centre PAUL STRAUSS, Strasbourg
- Germany (3):
  - University Hospital Dresden, Dresden
  - Asklepios Klinik Altona, Hamburg
  - Caritasklinikum Saarbruecken St Theresia, Saarbrücken
- Hungary (3):
  - Mav Korhaz Es Kozponti Rendelointezet, Budapest
  - Semmelweis Egyetem, Budapest
  - Clinexpert Kft Fázis I. Vizsgálóhely, Gyöngyös
- Italy (6):
  - AOU-S.Orsola-Malpighi - Universita degli Studi di Bologna, Bologna
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (IRST) IRCCS, Meldola
  - Instituto Europeo di Oncologia, Milan
  - Azienda Ospedaliero Universitaria Modena, Modena
  - Azienda Ospedaliero Universitaria Ospedali Riuniti Umberto I, Torrette
  - Ospedale Borgo Roma, Verona
- Portugal (3):
  - Hospital Senhora Da Oliveira - Hso-Epe, Guimarães
  - Centro Hospitalar Lisboa Norte - Hospital de Santa Maria, Lisbon
  - Fundacao Champalimaud, Lisbon
- Spain (14):
  - Chuac Hospital Teresa Herrera, A Coruña
  - Hospital Universitario de Badajoz, Badajoz
  - Hospital Universitario Vall D Hebron, Barcelona
  - Instituto Oncologico Dr Rosell Lor, Barcelona
  - Hospital Universitari de Lleida Arnaud de Villanova, Lleida
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Hospital Universitario Quiron Salud, Madrid
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Md Anserson Cancer Center, Madrid
  - Clinica Universidad de Navarra, Pamplona
  - Hospital Universitario Marques de Valdecilla, Santander
  - Complejo Hospitalario Universitario de Santiago de Compostela -Chus, Santiago de Compostela

IPD SHARING:
Plan to Share IPD: No